CLINICAL TRIAL: NCT04002882
Title: Outcomes Related to Body Composition in Teens and Adults With Cystic Fibrosis (ORBIT-CF)
Brief Title: Role of Body Fat Distribution in Metabolic and Pulmonary Decline in Cystic Fibrosis (ORBIT-CF)
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Jessica Alvarez, Assitant professor, Emory University
Other Study IDs: IRB00110358
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens that remain after completion of the study will be stored for future studies beyond the scope of the current study only if subjects denote the appropriate section of the informed consent form to grant long term storage of samples. Specimens and data will be stored at Emory University within the PI's (Jessica Alvarez) laboratory. Any stored samples will be de-identified with a specific code whose identity can only be accessed by authorized study personnel appointed by the PI.
  During the conduct of the study, an individual participant can choose to withdraw consent to have biological specimens stored for future research. However, withdrawal of consent with regard to bio-sample storage may not be possible after the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Subjects with Cystic Fibrosis: n=60 patients with CF ages 16-30
- Healthy Controls: n=30 healthy controls matched to participants with CF for age, sex, BMI, and race.

SUMMARY:
Nutrition and body composition, the amount of muscle and fat in the body, has a role in overall health. This study wants to learn more about how nutrition and body composition affects health outcomes like glucose tolerance and lung function in patients with cystic fibrosis (CF) who are ages 16-30 years old. 60 adolescents and young adults with CF will be recruited, and 30 volunteers without cystic fibrosis. A total of 40 of these study participants with CF will be asked to return for annual study visits for 2 years after the first visit.

The long-term goal of this study is to use the information collected to make decisions about future nutrition monitoring and interventions which help maintain optimal health for individuals with CF.

DETAILED DESCRIPTION:
This is a prospective, observation study to test the central hypothesis that individuals with cystic fibrosis (CF) have a higher propensity to increased visceral adipose tissue (VAT) accumulation and decreased lean body mass (LBM) compared to healthy controls, and this dysregulation in adipose and protein deposition exacerbates glucose intolerance and lung function decline. A sub-set of participants with CF will be followed longitudinally for two years (n=40). The investigators will conduct detailed body composition, fat distribution, metabolic, and nutritional phenotyping in this cohort. Body fat distribution will be assessed with MRI. Whole body composition will be assessed with DEXA. Glucose tolerance will be assessed with an oral glucose tolerance test (OGTT) and mathematical modeling of the C-peptide and insulin response to glucose. Lung health will be assessed by objective clinical data and self-reported symptoms.

ELIGIBILITY:
Inclusion Criteria:

CF inclusion criteria

1. confirmed CF diagnosis based on sweat testing by pilocarpine iontophoresis and/or CFTR genotyping with two disease causing mutations
2. be aged ≥ 16 yrs
3. clinically stable, defined as no changes in medical regimen (including medications) for at least 21 days prior to study visit
4. participation in the CFF Patient Registry

Longitudinal study inclusion:

CF participants who have normal glucose tolerance results after their initial study oral glucose tolerance test (OGTT).

Healthy controls inclusion criteria:

1. male or female ages 16 years and older
2. clinically stable. Healthy controls will be recruited who are similar in age, gender, and BMI as the participants with CF.

Exclusion Criteria:

CF exclusion criteria:

1. diagnosis of CF-related diabetes (CFRD)
2. nocturnal tube feeds
3. life expectancy <6 months
4. history of or on waiting list for lung transplant
5. un-removable metal that is incompatible with MRI
6. inability or unwillingness to perform major study activities (OGTT, DEXA, MRI) due to claustrophobia, fear of blood draw, or other reasons
7. current pregnancy or lactation
8. study visit falls between window of 1 week to 8 weeks of initiation of CFTR modulator
9. use of chronic oral corticosteroids,
10. in the opinion of the CF Care Team or study physician, participant should not participate in the study, or
11. inability to provide informed consent or assent.

Healthy controls exclusion criteria:

1. malignant neoplasm (other than localized basal cell cancer of the skin) during the previous 5 years
2. respiratory (including asthma), endocrine (including diabetes), autoimmune, or other chronic disease
3. HIV or other chronic infection
4. current use of any medications to treat an acute or chronic disease or illness (anti-depressants, anti-anxiety medications are acceptable),
5. acute illness within the past 3 weeks
6. intravenous or oral antibiotics or use of systemic corticosteroids within the past 3 weeks
7. inability or unwillingness to perform major study activities due to claustrophobia, fear of blood draw, or other reasons
8. current pregnancy or lactation, or
9. inability to provide informed consent or assent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This will be a two-site study of n=60 patients with CF ages 16 years and older and n=30 age-, sex-, BMI-, and race-matched healthy controls. As a sub-study, 40 of these CF subjects will be followed longitudinally and assessed annually for two years.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Visceral Adipose Tissue volume (VAT) by Magnetic Resonance Imaging (MRI) | Baseline, 1 year, 2 year
  Body fat distribution and body composition in 60 individuals with Cystic Fibrosis (CF) and 30 matched, healthy control will be assessed by Magnetic Resonance Imaging (MRI)
Change in Disposition Index | Baseline, 1 year, 2 year
  The disposition index (DI) is a measure of the ability of B-cells to compensate for insulin resistance.
  A lower DI indicates a loss of B-cell function, which means decreased pancreatic function. The disposition index will be assessed with an oral glucose tolerance test (OGTT) and mathematical modeling of the C-peptide and insulin response to glucose.
  This study seeks to determine if glucose intolerance is associated with body composition and fat distribution in CF subjects.
Change in Forced Expiratory Volume in the first second (FEV1%) | Baseline, 1 year, 2 year
  Clinical spirometry is a test of lung function that will be used to assess the progression of lung disease with the baseline Forced Expiratory Volume (FEV%) predicted within the past year. Baseline is defined as the average of the best FEV1% for each quarter of the calendar year. FEV1% predicted is a method of determining the severity of pulmonary disease and declines as disease severity increases.

SECONDARY OUTCOMES:
Change in Pancreatic lipid | Baseline, 1 year, 2 year
  Pancreatic lipid contributes to the Visceral Adipose Tissue volume (VAT) and it will me measured with the magnetic resonance imaging (MRI).
  Participants will lay in the supine position for approximately 30 minutes while in the MRI scanner, and images of the abdominal area (L1-L5 vertebrae) and thigh area will be obtained. Images will later be analyzed for quantification of VAT volume and lipid content of pancreas will be analyzed
Change in Hepatic lipid | Baseline, 1 year, 2 year
  Hepatic lipid contributes to the Visceral Adipose Tissue volume (VAT) and it will me measured with the MRI.
  Participants will lay in the supine position for approximately 30 minutes while in the MRI scanner, and images of the abdominal area (L1-L5 vertebrae) and thigh area will be obtained. Images will later be analyzed for quantification of VAT volume and lipid content of liver will be analyzed
Change in Thigh perimuscular adipose tissue (PMAT) | Baseline, 1 year, 2 year
  Thigh PMAT contributes to the VAT and it will me measured with the MRI. Participants will lay in the supine position for approximately 30 minutes while in the MRI scanner, and images of the abdominal area (L1-L5 vertebrae) and thigh area will be obtained. Images will later be analyzed for quantification of VAT volume and Thigh PMAT
Change in Body Composition Analysis | Baseline, 1 year, 2 year
  Dual-energy X-ray absorptiometry (DEXA) is an imaging technique that provides whole body and regional estimates of the three main body components: fat, lean soft tissues and bone mineral mass.
Change in Insulin secretion | Baseline, 1 year, 2 year
  Insulin secretion measures the total beta cell response (PhiTot), and will be assessed with an oral glucose tolerance test (OGTT).
  Fasted blood samples will be drawn 30 minutes and 15 minutes before the initiation of glucose consumption. At time "zero", an oral glucose solution at the dose of 1.75 gm/kg to a maximum of 75 gms will be provided and consumed within 5 minutes of administration. Subsequent blood samples will be drawn at 10, 20, 30, 60, 90, and 120 min following initiation of glucose ingestion.
  Decreased insulin secretion has been associated with lower B-cell function.
Change in Whole body insulin sensitivity index (WBISI) | Baseline, 1 year, 2 year
  Insulin sensitivity describes how sensitive the body is to the effects of insulin. Whole body insulin sensitivity index (WBISI) is derived from glucose and insulin levels from the full length of the OGTT. The index is calculated using a formula.
  Decreased insulin sensitivity index is associated with more advanced CF disease.
Annual rate of Forced Expiratory Volume in the first second (FEV1%) decline | Baseline, 1 year, 2 year
  FEV1 is the maximal amount of air you can forcefully exhale in one second. It is then converted to a percentage of normal, based on your height, weight, and race.
  It is assessed when doing the spirometry.
Number of pulmonary exacerbations needing intravenous (IV) antibiotics within previous five years | Baseline
  Number of pulmonary exacerbations needing intravenous (IV) antibiotics within previous five years will be recorded.
Number of Perceived respiratory symptoms measured with the Cystic Fibrosis Questionnaire-Revised (CFQ-R) | Baseline, 1 year, 2 year
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a disease-specific instrument, designed to measure impact on overall health, daily life, perceived well-being and symptoms.
  Scores range from 0 to 100, with higher scores indicating better health.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Alvarez, PhD, RD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - University of Alabama at Birmingham (UAB)/Children's of Alabama, Birmingham, Alabama
  - Emory University/Children's Hospital of Atlanta (CHOA), Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Completely de-identified participant data will be shared after publication of all results.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months following publication of results. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal that is approved by all primary study co-investigators.
  Types of analyses: To achieve the aims in the approved proposal and for individual participant data-meta analysis.
  Proposals should be directed to Dr. Alvarez at jessica.alvarez@emory.edu